CLINICAL TRIAL: NCT00849706
Title: Effect of Work Load and Sleep Deprivation on Medical Staff's Driving Skills
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Adar Tomer, Hadassah Medical Organization
Other Study IDs: 481131-HMO-CTIL
Record Dates: First submitted 2009-02-19; First posted 2009-02-24 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Sleep Deprivation
Keywords: sleep deprivation; workload; increased workload
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Study group: Medical staff personal, doctors and nurses, working night shifts.
  Interventions: Other: Study participants will work their regular shifts, and tested after night shifts.No shifts will be added because of the study.

INTERVENTIONS:
Other: Study participants will work their regular shifts, and tested after night shifts.No shifts will be added because of the study. — Night shifts in our medical center are working 8 hours from 23:00 to 7:00 the following day for nurses, and working overnight (24h) for doctors.

SUMMARY:
Long and unorthodox working hours (e.g. 24 hours or 23pm-07am shifts for doctors and nurses respectively) combined with sleep deprivation, may affect cognitive functions such as response time and concentration. These parameters may be tested using a driving simulator. Apart from the obvious consequences of driving skills impairment for the medical personal, it may serve as a quality assessment tool in evaluating the impact of workload and sleep deprivation on medical staff's function. This study aims to assess the effect of work load and sleep deprivation on medical staff's driving skills.

DETAILED DESCRIPTION:
Medical staff in Israel has long and unorthodox working hours. During residency, doctors stay overnight for shifts after working the normal working hours for a total of 24h, without regular set breaks or certainty of even one hour of sleep. Nurses, has three 8 hours shifts, changing at 7am, 3pm and 11pm, meaning the night shift staff works between 11pm and 7am the following morning. These conditions, especially when in a routine when one shifts follow another, may contribute to an accumulated workload, associated with sleep deprivation. Such conditions may have considerable impact on cognitive functions such as response time and concentration, which are fundamental for medical personal's function.

The driving simulator is based on software (STIS Drive Simulation software, System Technology INC, Hawthorne CA) and a hardware consisting of a computer, screen, and two consoles, one includes a stirring wheel and press buttons, the second includes acceleration and break paddles. Each test drive has several stages, in which the following are measured - the ability to maintain constant speed, the ability to maintain driving lain, to follow another vehicle and to break abruptly. Additionally, during the test drive, several arrows appear on the screen, and the subject is requested to push curtain buttons as they appear according to their direction. This simulator has been used in several prior reports for driving skills evaluation.

In this study, medical staff will be asked to be tested with the driving simulator after night shift, allowing assessment of cognitive functions and response time.

* Study design:

  * The study will include doctors and nurses from the internal medicine, surgical, orthopedic and pediatric wards which work night shifts.
  * The study will include both genders, ages 25-50.
  * The study is planned to include 100 volunteers.
* Trial entry and enrollment

  * The medical staff at the participating departments will be approached orally (staff meetings etc') and signs will be posted at staff rooms.
  * Willing volunteers will be enrolled according to order of consent.

    **Visits 1 and 2
  * Visit 1 will include a training session in which the volunteer is introduced to the driving simulator's different functions and will perform a test ride to get experience. At this session, the subject will be asked to fill a form stating his age, residency and main occupation (e.g. extent of familiarity with laparoscopic/ endoscopic procedures).
  * Visit 2 will include a test ride performed during morning (07:00- 14:00pm) and after a regular night sleep and not after a night shift. Data collected during this session will be considered as baseline values. The following three test visits will be compared to these values.

    ** Visits 3-5
  * These visits will be performed after night shifts. Subjects will be tested at the morning (7-10am) following a night shift. Apart form a test drive each subject will be asked to state work and sleep hour during the previous day.

    ** Visit 6
  * Subjects which have completed 3 test drives will undergo a repeat baseline assessment (similar to visit 2) to which the following visits will be compared in order to minimize the learning curve component.

    ** Visits 7-9
  * Similar to visits 3-5.
* Statistical considerations

  * Subjects will be grouped according to sleep hours prior to test drives, and driving simulator results will be compared.
  * Furthermore, additional analysis will be performed for individual subjects comparing achievements with sleep hours.
* Informed consent

  * Each subject will be enrolled and enter the study only after giving an informed consent.
* Adherence to study eligibility

  * The study will be conducted in accordance with good clinical practice (GCP) guidelines, and the study protocol.
* Safeguarding of documents

  * The privacy of the subjects and all confidentiality issues will be handled in accordance with applicable law and guidelines of the institution and the Helsinki Committee, the Israeli ministry of health, or the other appropriate regulatory authorities.

ELIGIBILITY:
Inclusion Criteria:

* Given informed consent
* Medical staff (doctor / nurse) working night shifts.
* Having a driver's license.

Exclusion Criteria:

* Pregnancy.
* Any systemic / neurological condition which may affect results.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Medical staff (doctors and nurses) working night shifts.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Change in driving simulator test results after night shifts compared with control. | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Ein-Kerem, Israel

REFERENCES:
- [Background] Bajaj JS, Hafeezullah M, Hoffmann RG, Varma RR, Franco J, Binion DG, Hammeke TA, Saeian K. Navigation skill impairment: Another dimension of the driving difficulties in minimal hepatic encephalopathy. Hepatology. 2008 Feb;47(2):596-604. doi: 10.1002/hep.22032. PMID 18000989
- [Background] Horne J, Reyner L. Vehicle accidents related to sleep: a review. Occup Environ Med. 1999 May;56(5):289-94. doi: 10.1136/oem.56.5.289. PMID 10472301